CLINICAL TRIAL: NCT01174225
Title: Contraception Satisfaction and Effectiveness: A Randomized Controlled Trial
Brief Title: IUD Insertion Post First Trimester Abortion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Wendy Norman, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H10-00798
Record Dates: First submitted 2010-07-30; First posted 2010-08-03 (Estimated); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Contraception
Keywords: Copper IUD; Nova T 200; Flexi T 380; expulsion; contraception satisfaction; post-abortion contraception
MeSH Terms: interventions — Intrauterine Devices

STUDY DESIGN:
Intervention Model Description: Flexi-T380(+) IUD Nova-T200 IUD
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- I (Active Comparator): Participants who elect to have an IUD inserted at the time of abortion will be randomized to either Arm I or Arm II. In this arm participants will receive the Flexi T 380(+) IUD. The participant is counseled that she may leave the device in for up to five years. She will be followed for up to five years to determine expulsion rate, discontinuation rate, pregnancy rate, and overall satisfaction with form of contraception.
  Interventions: Device: Flexi T 380(+) IUD
- II (Active Comparator): Participants who elect to have an IUD inserted at the time of abortion will be randomized to either Arm I or Arm II. In this arm participants will receive the Nova T IUD. The participant is counseled that she may leave the device in for up to five years. She will be followed for up to five years to determine expulsion rate, discontinuation rate, pregnancy rate, and overall satisfaction with form of contraception.
  Interventions: Device: Nova T IUD
- III (No Intervention): Participants who elect for forms of contraception other than a copper IUD will chose which form of contraception they would like to use and be put into one of the groups specified below based on her contraceptive choice. These participants will be observed throughout the study for overall satisfaction and repeat pregnancy rate.
  Groups - Participants will be in one of the five following groups Group A - Oral contraceptive pill 28day supply provided after abortion Group B - Medroxyprogesterone acetate (Depo-provera)150mg IM provided after abortion, lasts for 3 months Group C - Ethinyl estradiol and etonogestrel (Nuva ring) provided at time of abortion, lasts for 28 days Group D - Condoms provided at time of abortion Group E - Other

INTERVENTIONS:
Device: Flexi T 380(+) IUD — The intrauterine device is placed in the uterus immediately post-abortion. Participant is counseled that she may leave the device in for up to five years.
  Arms: I
Device: Nova T IUD — The intrauterine device is placed in the uterus immediately post-abortion. Participant is counseled that she may leave the device in for up to five years.
  Arms: II

SUMMARY:
The goal of this study is to provide better information about contraception to women having an abortion so that they are less likely to have another unintended unwanted pregnancy.

Participating subjects will receive their choice of contraception following their abortion and if this choice is an IUD they will be randomly assigned to one of two types of copper intrauterine devices.

All participating women will fill out a survey about their contraceptive choices at the time of their abortion as well as at 3, 6, and 12 months afterwards. The investigators will also follow pregnancy rates at 1 through 5 years after the abortion to see which form of contraception was most effective.

The investigators expect to find that IUDs are the most effective form of contraception but that the types of copper IUDs currently available in Canada are not known to be as effective as those available in other countries, for which high quality evidence is available. The investigators hope to use this data to determine the effectiveness of copper IUDs available in Canada.

DETAILED DESCRIPTION:
This prospective randomized controlled trial will examine satisfaction and effectiveness of post abortion contraception by comparing the two types of copper IUDs currently available in Canada, and including a non-interventional group of other contraceptive options.

The primary outcome measure is one year expulsion rates of copper IUDs places post abortion. Secondary outcomes are satisfaction with current method at 3, 6, and 12 months post-abortion, retention rates and repeat abortion rate over one year. One and five year pregnancy rates will be analyzed using access to universal health care databases.

Our results will provide the first information on the effectiveness of post abortion contraceptive methods currently available in Canada.

ELIGIBILITY:
Inclusion Criteria:

* Residents of BC registered with the Medical Services Plan of British Columbia
* Women seeking abortions for pregnancies up to 11 weeks 6 days gestation

Key Exclusion Criteria:

* Women who plan to conceive within the next year

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 534 (Actual)
Dates: Start 2010-09; Primary Completion 2013-09 (Actual); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
The expulsion rate of each IUD | 12 months
  The expulsion rate of each IUD and the scaled measure of patient satisfaction with each form of contraception (completed July 2012)

SECONDARY OUTCOMES:
Voluntary discontinuation rate of contraception | 12 months
  Voluntary discontinuation rate of contraception and one year rates of repeat abortion (completed July 2012)
  - One and five year pregnancy rate for each form of contraception chosen (completed 2018)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy V Norman, MD, FCFP, Principal Investigator — University of British Columbia
Locations (1):
- Kelowna Womens' Clinic, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Samiedaluie S, Peterson S, Brant R, Kaczorowski J, Norman WV. Validating abortion procedure coding in Canadian administrative databases. BMC Health Serv Res. 2016 Jul 12;16:255. doi: 10.1186/s12913-016-1485-4. PMID 27406214
- [Derived] Norman WV, Chiles JL, Turner CA, Brant R, Aslan A, Kaczorowski J. Comparing the effectiveness of copper intrauterine devices available in Canada. Is FlexiT non-inferior to NovaT when inserted immediately after first-trimester abortion? Study protocol for a randomized controlled trial. Trials. 2012 Aug 24;13:147. doi: 10.1186/1745-6215-13-147. PMID 22920273
- See also: This website is the site for the Research Team and summarizes current studies — http://www.cart-grac.ubc.ca